CLINICAL TRIAL: NCT06512688
Title: Establishing Reference Ranges for Fat-Soluble Vitamins in Healthy Chinese Adults
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Huizhou Municipal Central Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Zhejiang Provincial Tongde Hospital (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Zhejiang Provincial People's Hospital (Other); Affiliated Hangzhou First People's Hospital (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); Lu'an People's Hospital of Anhui Province (Unknown); Shandong Provincial Hospital (Other Government); Second Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Nanchang University (Other); Nanfang Hospital, Southern Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Changzhi Medical College (Other); LinFen People's Hospital (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Yulin No.2 Hospital (Other); Hanzhong Central Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhong, Head of Health Management Center, First Affiliated Hospital of Zhejiang University
Other Study IDs: 20240364
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Fat Soluble Vitamin Deficiencies and Disorders
Keywords: Reference Interval; Healthy Chinese Adults
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — This is a cross-sectional study without intervention.

SUMMARY:
Vitamins are essential micronutrients required for maintaining normal physiological functions and metabolism in humans. Among them, fat-soluble vitamins (FSV) such as vitamins A, D, E, and K are absorbed in the intestines in the presence of fat. Both deficiencies and excesses of these vitamins can affect health. Current global studies on FSVs in healthy populations are often limited to specific types or regions, and comprehensive data on all four FSVs in the healthy Chinese population are lacking. This study aims to fill this gap by collecting and analyzing FSV levels from healthy adults across multiple regions in China, establishing a reference range for clinical evaluation and early disease intervention.

DETAILED DESCRIPTION:
Vitamins are crucial organic micronutrients necessary for maintaining human physiological functions and metabolic processes. They are typically categorized into water-soluble vitamins and fat-soluble vitamins (FSVs). The primary FSVs include vitamins A, D, E, and K, which are absorbed in the intestines in the presence of dietary fat.

The balance of these vitamins in the body is vital for health. Deficiencies or excesses can lead to significant health issues. For example, a deficiency in vitamin A can cause night blindness, a lack of vitamin D can lead to osteomalacia, insufficient vitamin E can result in increased oxidative stress in cells, and a deficiency in vitamin K can cause bleeding disorders.

Globally, research on FSVs in healthy populations is usually focused on specific vitamins or limited to particular regions and demographics. Consequently, there is a scarcity of comprehensive data on the concentration of all four FSVs at the population level. In China, there has been no extensive study that simultaneously analyzes the levels of all four FSVs in a healthy adult population.

This study addresses this gap through a multicenter approach, collecting data on the levels of vitamins A, D, E, and K from healthy adults across various regions in China. The goal is to establish a reference range for serum FSV levels in Chinese adults. This database will serve as a scientific foundation for accurately assessing FSV levels in clinical settings and providing early intervention for diseases related to FSV imbalances. Additionally, this research aims to enhance understanding of the nutritional status of the Chinese population and guide dietary recommendations and public health policies to improve overall health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, both male and female;
2. Undergo a health examination in this hospital and consciously maintain good physical health;
3. Voluntarily participate in this study and sign an informed consent form;
4. No acute and chronic diseases: no acute and chronic infections, cardiovascular and cerebrovascular diseases, diabetes, respiratory diseases, urinary diseases, thyroid diseases, digestive diseases, rheumatic diseases, blood system diseases, tumors, pituitary dysfunction; No hepatitis B, hepatitis C virus, or acquired immunodeficiency syndrome;
5. Blood pressure: systolic blood pressure<140 mmHg and diastolic blood pressure<90 mmHg;
6. BMI (body mass index):<28 kg/m2 and ≥ 18.5 kg/m2;
7. No surgery was performed within 6 months, no blood donation, transfusion, or significant blood loss occurred within 4 months;
8. No long-term medication history, no medication or vitamin supplements taken within 2 weeks;
9. Women who are not pregnant, breastfeeding, or within one year after childbirth;
10. No alcohol abuse (alcohol consumption but alcohol intake<140 g/week for males and<70 g/week for females), and smoking (<20 cigarettes/day).

Exclusion Criteria:

1. Serum alanine aminotransferase (ALT): Male>50 U/L, female>40 U/L; Or serum gamma glutamyltransferase (GGT): male>60 U/L, female>45 U/L; Or serum aspartate aminotransferase (AST): male>40 U/L, female>35 U/L; Or serum alkaline phosphatase (ALP): male>125 U/L, female (20-49 years old)>100 U/L, female (50-79 years old)>100 U/L;
2. Serum albumin (ALB) < 40 g/L;
3. Serum creatinine (SCr): Male (20-59 years old)>97 μ mol/L, male (60-79 years old)>111 μ mol/L; Female (20-59 years old)>73 μ mol/L, female (60-79 years old)>81 μ mol/L;
4. Fasting blood glucose (FBG) ≥ 7.0 mmol/L;
5. White blood cell count (WBC): < 3.5 × 109/L or > 9.5 × 109/L;
6. Hemoglobin (Hb): Male < 120 g/L; Female<110 g/L;
7. Glycated hemoglobin (HbA1c)<4% or>6%;
8. Total cholesterol (TC) ≥ 5.2 mmol/L; Or triglycerides (TG) ≥ 1.7 mmol/L;
9. Low density lipoprotein cholesterol (LDL-C) ≥ 3.4 mmol/L; Or high-density lipoprotein cholesterol (HDL-C)<1.0 mmol/L;
10. Serum uric acid (UA)>420 μ mol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and above who underwent physical examinations in collaborating hospitals from July 2024 to June 2026.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
serum vitamin A | day 1
serum vitamin D | day 1
serum vitamin E | day 1
serum vitamin K | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Liu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No